CLINICAL TRIAL: NCT04371666
Title: A Phase 3, Randomized, Double-Blind Trial of Pamrevlumab (FG-3019) or Placebo in Combination With Systemic Corticosteroids in Subjects With Non-ambulatory Duchenne Muscular Dystrophy (DMD)
Brief Title: Phase 3 Trial of Pamrevlumab or Placebo With Systemic Corticosteroids in Participants With Non-ambulatory Duchenne Muscular Dystrophy (DMD)
Acronym: LELANTOS-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study did not meet its primary endpoint.
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-3019-093; 2020-000698-26 (EudraCT Number)
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy, DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — pamrevlumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pamrevlumab (Experimental): Pamrevlumab 35 milligrams (mg)/kilogram (kg) intravenously (IV) every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks
  Interventions: Drug: Pamrevlumab; Drug: Corticosteroids
- Placebo (Placebo Comparator): Matching placebo IV every 2 weeks + systemic deflazacort or equivalent potency of corticosteroids administered orally for up to 52 weeks
  Interventions: Drug: Placebo; Drug: Corticosteroids

INTERVENTIONS:
Drug: Pamrevlumab — Pamrevlumab per dose and schedule specified in the arm description
  Other Names: FG-3019
  Arms: Pamrevlumab
Drug: Placebo — Matching placebo per schedule specified in the arm description
  Arms: Placebo
Drug: Corticosteroids — Systemic deflazacort or equivalent potency of corticosteroids administered orally

SUMMARY:
To evaluate the efficacy and safety of pamrevlumab versus placebo in combination with systemic corticosteroids in participants with non-ambulatory Duchenne muscular dystrophy (age 12 years and older).

DETAILED DESCRIPTION:
This is a global, Phase 3, randomized, double-blind trial of pamrevlumab or placebo in combination with systemic corticosteroids in participants with non-ambulatory Duchenne muscular dystrophy, aged 12 years and older. Approximately 90 male participants will be randomized at a 1:1 ratio to Arm A (pamrevlumab + systemic corticosteroid) or Arm B (placebo+ systemic corticosteroid), respectively.

Participants must be fully informed of the potential benefits of approved products and make an informed decision that they prefer to participate in a clinical trial in which they could be randomized to placebo.

This trial has 3 study periods:

* Screening period: Up to 4 weeks
* Treatment period: 52 weeks
* Safety Follow-up period/End of Study (EOS): A visit 28 days (+/- 3 Days) and a final safety follow-up phone call 60 days (+ 3 Days) after the last dose

In the screening period, participants will be evaluated per the protocol inclusion/exclusion criteria to determine eligibility for participation in this trial.

During the treatment period, each participant will receive pamrevlumab or placebo at 35 mg/kg every 2 weeks for up to 52 weeks.

Participants who complete the 52-week study (either arm) may be eligible for rollover into an open-label extension treatment (OLE) with pamrevlumab + systemic corticosteroids.

Participants who discontinue study treatment for any reason should be encouraged to return to the investigative site to complete final safety and efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Males at least 12 years of age, non-ambulatory at screening initiation
2. Written consent by participant and/or legal guardian as per regional/ country and/or Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements
3. Male participants with partners of childbearing potential must use contraception during the conduct of the study, and for 12 weeks after the last dose of study drug.
4. Medical history includes diagnosis of DMD and confirmed Duchenne mutation using a validated genetic test
5. Brooke Score for Arms and Shoulders ≤5
6. Able to undergo MRI test for the upper arm extremities (Biceps Brachii muscle) and cardiac muscle
7. Able to perform spirometry
8. Average (of Screening and Day 0) percent predicted forced vital capacity (FVC) between 45 and 85, inclusive
9. Left ventricular ejection fraction ≥50% as determined by local cardiac MRI read at screening or within 3 months prior to randomization (Day 0)
10. If participants have a history of cardiomyopathy, then participant must be on a stable dose of cardiomyopathy/ heart failure medications (for example, angiotensin converting enzyme inhibitors, aldosterone receptors blockers, angiotensin-receptor blockers, and betablockers) for at least 1 month prior to screening. If participants have no diagnosis of cardiomyopathy, then no dose of cardiomyopathy/heart failure medication is required for eligibility.
11. On a stable dose of systemic corticosteroids for a minimum of 6 months, with no substantial change in dosage for a minimum of 3 months (except for adjustments for changes in body weight) prior to screening. Corticosteroid dosage should be in compliance with the DMD Care Considerations Working Group recommendations (for example, prednisone or prednisolone 0.75 mg/kg per day or deflazacort 0.9 mg/kg per day) or stable dose. A reasonable expectation is that dosage and dosing regimen would not change significantly for the duration of the study.
12. Agreement to receive annual influenza vaccinations during the course of the study.
13. Adequate renal function: cystatin C ≤1.4 mg/liter (L)
14. Adequate hematology and electrolytes parameters:

    1. Platelets >100,000/microliter (μL)
    2. Hemoglobin >12 grams (g)/deciliter (dL)
    3. Absolute neutrophil count >1500/μL
    4. Serum calcium (Ca), potassium (K), sodium (Na), magnesium (Mg) and phosphorus (P) levels are within a clinically accepted range for DMD participants.
15. Adequate hepatic function:

    1. No history or evidence of liver disease
    2. Gamma glutamyl transferase (GGT) ≤3x upper limit of normal (ULN)
    3. Total bilirubin ≤1.5xULN

Exclusion Criteria:

1. Previous exposure to pamrevlumab
2. BMI ≥40 kg/square meter (m^2) or weight >117 kg
3. History of:

   1. allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies
   2. hypersensitivity to study drug or any component of study drug
   3. hypersensitivity reaction to Gadolinium-based Contrast Agents (GBCA) required for MRI acquisition
4. Exposure to any investigational drug (for DMD or not), in the 30 days prior to screening initiation or use of approved DMD therapies (for example, eteplirsen [exondys 51], ataluren, golodirsen [vyondys 53], casimersen [amondys 45]) within 5 half-lives of screening, whichever is longer, with the exception of the systemic corticosteroids, including deflazacort
5. Severe uncontrolled heart failure (NYHA Classes III-IV), or renal dysfunction, including any of the following:

   1. Need for intravenous diuretics or inotropic support within 8 weeks prior to screening
   2. Hospitalization for a heart failure exacerbation or arrhythmia within 8 weeks prior to screening
   3. Participants with glomerular filtration rate (GFR) of less than 30 mL/minute (min)/1.73 m^2 or with other evidence of acute kidney injury as determined by investigator
6. Arrhythmia requiring anti-arrhythmic therapy
7. Requires ≥16 hours continuous ventilation
8. Hospitalization due to respiratory failure within the 8 weeks prior to screening
9. Poorly controlled asthma or underlying lung disease such as bronchitis, bronchiectasis, emphysema, recurrent pneumonia that in the opinion of the investigator might impact respiratory function
10. The Investigator judges that the participant will be unable to fully participate in the study and complete it for any reason, including inability to comply with study procedures and treatment, or any other relevant medical or psychiatric conditions

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (24):
  - Arkansas Children's, Little Rock, Arkansas
  - University of California Los Angeles Medical Center, Los Angeles, California
  - UC Davis Health, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Fairway, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - UMASS Med School, Worcester, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Spectrum Health Hospitals Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Washington University School of Medicine in Saint Louis, St Louis, Missouri
  - Carolinas HealthCare System Neurosciences Institute-Neurology - Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Shriners Hospital for Children, Portland, Oregon
  - Penn State Health Children's Hospital, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Health Dallas/UTSW, Dallas, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Children's Specialty Group - Medical Center Office, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Klinik Favoriten, Vienna, Austria
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Régional de la Citadelle, Liège
- London Health Sciences Centre, London, Ontario, Canada
- China (3):
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
- Czechia (2):
  - Fakultní Nemocnice Brno - Dětská Nemocnice, Brno
  - Klinika dÄ>tské neurologie, Neuromuskulární centrum, Prague
- France (3):
  - CHU de Nantes - Hotel Dieu, Nantes
  - Association Institut de Myologie, Paris
  - Hopital Hautepierre, Strasbourg
- Israel (2):
  - The Chaim Sheba Medical Center, Tel Aviv
  - The Edith Wolfson Medical Center, Tel Aviv
- Italy (4):
  - Istituto di Ricovero e Cura a Carattere Scientifico Eugenio Medea - Lombardia, Lecco
  - IRRCS Ospedale San Raffaele, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome
  - Ospedale Pediatrico Bambino Gesù - Roma - Gianicolo, Rome
- Netherlands (2):
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Leiden Universitair Medisch Centrum, Leiden
- Spain (3):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- Inselspital Universitätsspital Bern, Bern, Switzerland
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University College London Hospitals NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included 2 periods: Double-blind (DB) Treatment Period and Open-label Extension (OLE) Period.
Groups:
- Pamrevlumab: Participants received pamrevlumab intravenously (IV) every 2 weeks for up to 52 weeks in the DB treatment period. After completing Week 52 of the DB treatment period, participants in the OLE period then moved to Week 2 of the OLE period and received pamrevlumab IV every 2 weeks.
- Placebo: Participants received placebo matched to pamrevlumab IV every 2 weeks for up to 52 weeks in the DB treatment period. After completing Week 52 of the DB treatment period, participants in the OLE period then moved to Week 2 of the OLE period and received pamrevlumab IV every 2 weeks.
Period: DB Treatment Period (52 Weeks)
Arm/Group | Pamrevlumab | Placebo
Started | 49 | 49
Received at Least 1 Dose of Study Drug | 48 | 49
Completed | 44 | 46
Not Completed | 5 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Participant/Legal Guardian Decision | 1 | 2
Not completed — Other than specified | 1 | 0
Period: OLE (Maximum Exposure: 93.4 Weeks)
Arm/Group | Pamrevlumab | Placebo
Started | 43 | 43
Received at Least 1 Dose of Study Drug | 43 | 43
Completed | 0 | 0
Not Completed | 43 | 43
Not completed — Participant/Legal Guardian Decision | 2 | 2
Not completed — Sponsor Decision to Terminate Study | 40 | 41
Not completed — Other than specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) set included all randomized participants.
Groups:
- Pamrevlumab: Participants received pamrevlumab IV every 2 weeks for up to 52 weeks in the DB treatment period. After completing Week 52 of the DB treatment period, participants in the OLE period then moved to Week 2 of the OLE period and received pamrevlumab IV every 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Pamrevlumab | Placebo | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (2.74) | 15.5 (2.42) | 15.5 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 49 | 49 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 44 | 41 | 85
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 42 | 35 | 77
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Score of Performance of Upper Limb (PUL) 2.0 Version at Week 52
Description: The PUL module is an observer-administered performance battery of upper extremity mobility tasks for the shoulder (upper, 6 items, 12 points), elbow (middle, 9 items, 17 points) and wrist/hand (distal, 7 items, 13 points). Higher scores indicate higher level of function. Total score ranges from 0-42 points and is the sum of the scores for the 3 subscales. Analysis was done using a random coefficient model (RCM), which included fixed effects of time (as a continuous variable), treatment, and treatment-by-time interaction, with baseline ordinal PUL entry score as covariate.
Time Frame: Baseline, Week 52
Population: The modified intent-to-treat (mITT) population included all randomized participants with a PUL Entry score ≥2 (excluding PUL entry scores of 1) at baseline. Here, 'Overall number of participants analyzed' = participants evaluable for specified outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Pamrevlumab: Participants received pamrevlumab IV every 2 weeks for up to 52 weeks in the DB treatment period.
- Placebo: Participants received placebo matched to pamrevlumab IV every 2 weeks for up to 52 weeks in the DB treatment period.
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 38 | 40
units on a scale | -2.036 (0.4471) | -2.119 (0.3367)
Statistical Analysis 1: Comparison: Pamrevlumab vs Placebo; Test type: Other; p = 0.8802, Random coefficient model — Threshold for significance at 0.05 level; Least square (LS) Mean Difference = 0.083, 95% CI 2-sided [-1.010 to 1.176], Standard Error of Mean 0.5494

2. Secondary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (ppFVC) at Week 52, Assessed by Spirometry
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted FVC is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%. Analysis was done using an RCM, which included fixed effects of time (as a continuous variable), treatment, and treatment-by-time interaction, with baseline value as covariate.
Time Frame: Baseline, Week 52
Population: The mITT population included all randomized participants with a PUL Entry score ≥2 (excluding PUL entry scores of 1) at baseline. Here, 'Overall number of participants analyzed' = participants evaluable for specified outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted FVC
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 38 | 40
percentage of predicted FVC | -8.349 (1.5760) | -5.989 (1.2233)

3. Secondary Outcome: Change From Baseline in the Grip Strength of the Hands at Week 52, Assessed by Hand Held Myometry (HHM)
Description: The HHM was used to measure distal upper arm strength (grip strength). Data has been presented by dominant and non-dominant hand. Grip Strength was analyzed using a MMRM with fixed effects for treatment, visit (as a factor), treatment-by-visit interaction, and covariates (baseline values).
Time Frame: Baseline, Week 52
Population: The mITT population included all randomized participants with a PUL Entry score ≥2 (excluding PUL entry scores of 1) at baseline. Here, 'Overall number of participants analyzed' = participants evaluable for specified outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Least Squares Mean (Standard Error); unit: newton
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 37 | 39
newton
  Grip Strength by Dominant Hand | -7.570 (2.0989) | -0.072 (2.2065)
  Grip Strength by Nondominant Hand: number analyzed (Participants) | 36 | 39
  Grip Strength by Nondominant Hand | -7.627 (1.8893) | -0.012 (1.8546)

4. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction Percentage (LVEF %) at Week 52, Assessed by Magnetic Resonance Imaging (MRI)
Description: LVEF% is an important measure of cardiac function. LVEF is a fraction of blood (in percent) pumped out of the left ventricle of the heart (the main pumping chamber). The LVEF% was analyzed using an analysis of covariance (ANCOVA) model with treatment and baseline value.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of LVEF
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 33 | 37
percentage of LVEF | -0.499 (0.9750) | -1.114 (0.9204)

5. Secondary Outcome: Change From Baseline in Percent Predicted Peak Expiratory Flow (ppPEF) at Week 52, Assessed by Spirometry
Description: The ppPEF is a measure of the maximal or peak flow produced during an exhalation with maximal effort and, as such, is the most effort-dependent measure of lung function. The ppFEV1 was analyzed using an RCM including fixed effects of time, treatment, and treatment-by-time interaction, with baseline as covariate.
Time Frame: Baseline, Week 52
Population: The ITT set included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for specified outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted PEF
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 46 | 47
percentage of predicted PEF | -4.921 (2.3086) | -4.516 (1.7663)

ADVERSE EVENTS:
Time Frame: DB treatment period: From first dose of study drug up to 61 weeks OLE period: From first dose of study drug up to study termination by Sponsor and safety follow-up (up to approximately 102 weeks)
Description: The safety analysis set included all participants who received any dose of study medication.
Groups:
- DB Period: Pamrevlumab: Participants received pamrevlumab IV every 2 weeks for up to 52 weeks in the DB treatment period.
- DB Period: Placebo: Participants received placebo matched to pamrevlumab IV every 2 weeks for up to 52 weeks in the DB treatment period.
- OLE Period: Pamrevlumab: After completing Week 52 of the DB treatment period, participants in the OLE period then moved to Week 2 of the OLE period and received pamrevlumab IV every 2 weeks.
Arm/Group | DB Period: Pamrevlumab | DB Period: Placebo | OLE Period: Pamrevlumab
All-Cause Mortality (participants affected / at risk) | 1/48 | 0/49 | 0/86
Serious Adverse Events (participants affected / at risk) | 8/48 | 6/49 | 5/86
Other Adverse Events (participants affected / at risk) | 42/48 | 44/49 | 53/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Pamrevlumab (N=48) | DB Period: Placebo (N=49) | OLE Period: Pamrevlumab (N=86)
Myocarditis (Cardiac disorders) | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 3 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Testicular necrosis (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Pamrevlumab (N=48) | DB Period: Placebo (N=49) | OLE Period: Pamrevlumab (N=86)
Cardiomyopathy (Cardiac disorders) | 1 | 5 | 0
Cataract (Eye disorders) | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 10 | 5 | 5
Nausea (Gastrointestinal disorders) | 8 | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 4
Pyrexia (General disorders) | 12 | 4 | 14
Pain (General disorders) | 4 | 0 | 0
COVID-19 (Infections and infestations) | 19 | 19 | 10
Nasopharyngitis (Infections and infestations) | 3 | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 6 | 3 | 2
Rhinitis (Infections and infestations) | 1 | 4 | 4
Vascular access site bruising (Injury, poisoning and procedural complications) | 3 | 4 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 2 | 4
Limb injury (Injury, poisoning and procedural complications) | 4 | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 3 | 0
Heart rate increased (Investigations) | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Headache (Nervous system disorders) | 25 | 10 | 24
Dizziness (Nervous system disorders) | 4 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 0
Flushing (Vascular disorders) | 3 | 2 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Femur fracture (Injury, poisoning and procedural complications) | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT04371666/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT04371666/SAP_001.pdf